CLINICAL TRIAL: NCT02746692
Title: Faster Back Home: a Randomized Controlled Equivalence Study on the Efficacy of a High-intensity 15 Minute Aerobic Endurance Training
Brief Title: Faster Back Home: Efficacy of a High-intensity Endurance Training
Acronym: Fit15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SpM2016-003
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Fit15
- Comparison (Active Comparator)
  Interventions: Other: Endurance

INTERVENTIONS:
Other: Fit15 — Group-based high-intensity circuit training based on functional movement patterns (e.g. squats, push-ups, burpees, jumps, ropeskipping).
  Total duration 15 minutes circle training: 20s workout, 10 rest
  Arms: Intervention
Other: Endurance — Moderate intensity ergometer training. Total duration 50 minutes
  Arms: Comparison

SUMMARY:
Sports medical experts recommend considerable amounts of regular physical activity in order to improve strength, motor control, endurance and flexibility. However, only a small share of the population is able to meets the corresponding international guidelines. One reason for this is supposed to consist in private scheduling problems and the high time expenditure. Against this background, high-intensity intermittent training methods with short durations have become popular.

The present study aims to evaluate the effectivity of a high -intensity functional circuit training (the FIT15 program) in improving body function.

Thirty healthy individuals will be included in the randomized, controlled two-armed parallel group trial. In the intervention group, the participants will perform the FIT15 program, a group-based high-intensity circuit training based on functional movement patterns (e.g. squats, push-ups, burpees, jumps, rope-skipping). The training will be carried out three times a week, each 15 minutes for a total of six weeks. In the control group, the participants will exercise three times a week (in total for six weeks) at moderate intensity on an ergometer according to the cardiopulmonary exercise guidelines of the American College of Sports Medicine. Outcomes assess prior and following the six-week training period encompass body fat and muscle mass (bio impedance analysis), aerobic exercise capacity (spirometric exercise testing including lactate analysis), postural control (force plate), maximum strength of the leg extensors and shoulder muscles (1 repetition maximum) and psychometric variables (e.g. physical activity readiness questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* subscribing informed consent

Exclusion Criteria:

* Drug intake in the past 48 hours
* Pregnancy
* Muscle soreness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Maximal ventilatory aerobic endurance capacity assessed by spiroergometry | 10 min.
Maximal lactate aerobic endurance capacity assessed by spiroergometry | 10 min.

SECONDARY OUTCOMES:
Jumping performance; counter movement jump | 1 min.
Dynamic balance assessed with the time to stabilization test | 2 min
Static balance assessed with the time to stabilization test | 2 min
Maximal isometric voluntary force of the shoulder muscles | 10 min
Maximal isometric voluntary force of the lower limb extensors | 10 min
body composition assessed with a external non-invasive impedance device | 10 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany